CLINICAL TRIAL: NCT06752655
Title: The Effect of Photodynamic Therapy Using Curcumin As a Photosensitizer on Postoperative Pain After Non-Surgical Root Canal Retreatment: a Randomized Controlled Clinical Trial
Brief Title: Postoperative Pain in Photodynamic Therapy Using Curcumin As a Photosensitizer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Meltem Sümbüllü, Assistant Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 404380
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Periapical Diseases; Postoperative Dental Pain; Irrigation Solution; Photodynamic Therapy (PDT)
Keywords: postoperative pain; endodontics; root canal irrigation; curcumin; photodynamic therapy
MeSH Terms: conditions — Periapical Diseases; Pain, Postoperative | interventions — Curcumin; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curcumin with photodynamic therapy (Experimental): Root canal lengths will be determined using an electronic apex locator with a 15-K file. R25 and R50 Reciproc files will be used at working lengths to complete the canal preparation. During instrumentation, the root canals will be irrigated with 2 mL of 1% NaOCl. Subsequently, the root canals will be dried with paper points, and the final irrigation procedure will be performed using a curcumin solution in combination with photodynamic therapy. The root canals will then be filled with gutta-percha and sealer, and the coronal restoration will be completed. Patients will be provided with a form to assess postoperative pain and asked to score it daily. The completed form will be requested after one week.
  Interventions: Other: Curcumin with photodynamic thearpy
- control group (Active Comparator): Root canal lengths will be determined using an electronic apex locator with a 15-K file. R25 and R50 Reciproc files will be used at working lengths to remove the canal filling. During instrumentation, the root canals will be irrigated with 2 mL of NaOCl (1%). Subsequently, the root canals will be dried with paper points, and the final irrigation procedure will be performed using NaOCl (1%) and EDTA (17%) solutions. The root canals will then be filled with gutta-percha and sealer, and the coronal restoration will be completed. Patients will be provided with a form to assess postoperative pain and asked to score it daily. The completed form will be requested after one week.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Curcumin with photodynamic thearpy — root canals will irrigated with final irrigation procedure: curcumin+photodynamic therapy. The teeth will be isolated with a rubber dam, and an access cavity will be created. After root canal preparation, the final irrigation procedure will be performed. Root canal treatments will be completed, and the patients' postoperative pain levels will be recorded using follow-up forms.
  Arms: Curcumin with photodynamic therapy
Other: Control group — root canals will irrigated with routine root canal final irrigation with NaOCl and EDTA. The teeth will be isolated with a rubber dam, and an access cavity will be created. After root canal preparation, the final irrigation procedure will be performed. Root canal treatments will be completed, and the patients' postoperative pain levels will be recorded using follow-up forms.
  Arms: control group

SUMMARY:
In endodontics, various irrigation solutions are used to achieve antibacterial efficacy within the root canal. The antibacterial effect of curcumin-containing root canal solutions, when combined with photodynamic therapy, has been demonstrated in several studies. However, no research has specifically examined their effect on postoperative pain. The aim of this study is to investigate the impact of using a curcumin solution in combination with photodynamic therapy as the final irrigation solution on postoperative pain.

DETAILED DESCRIPTION:
Fifty patients were randomly assigned to two groups using a web-based program, according to the selected final irrigation procedure: curcumin-photodynamic therapy or a control group (routine root canal final irrigation with NaOCl and EDTA). The teeth will be isolated with a rubber dam, and access cavities will be created. After root canal preparation, the final irrigation procedure will be performed. Root canal treatments will then be completed, and the patients' postoperative pain levels will be recorded using follow-up forms.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients with aged between 18-60.
* Incisor, canine, and premolar teeth that had previously undergone root canal treatment
* Incisor, canine, and premolar teeth with a diagnosis of chronic apical abscess or asymptomatic apical periodontitis
* teeth with only 1 root canal
* the patients had not used any antibiotics for 3 months before treatment

Exclusion Criteria:

* the presence of a root fracture
* teeth with any swelling
* ankyloses,
* periodontal pockets deeper than 4 mm.
* teeth which a rubber dam could not be performed
* patients with allergy to ibuprofen or ciprofloxacin were also excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
postoperative pain levels | one week
  postoperative pain levels will be describe using the visual analog scale (VAS). The VAS was classified using the following scale [15]: no pain (0); mild pain (1-3); moderate pain (4-6), and severe pain (7-10).

SECONDARY OUTCOMES:
dependent variables-sex | one week
  The patients' genders (female or male) will be recorded, and their relationship with postoperative pain will be statistically analyzed.
dependent variable-age | one week
  The patients' ages will be recorded as numbers, and their relationship with postoperative pain will be statistically analyzed.
dependent variables-teeth number | one week
  The patients' tooth numbers will be recorded, and their relationship with postoperative pain will be statistically analyzed.
dependent variables-smoking habit | one week
  The patients' smoking habits will be recorded as either "yes" or "no," and their relationship with postoperative pain will be statistically analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Erzurum, yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No